CLINICAL TRIAL: NCT01227018
Title: Phase II Study of STA-9090 as Second or Third-Line Therapy for Metastatic Pancreas Cancer
Brief Title: PhII Study STA-9090 as Second or Third-Line Therapy for Metastatic Pancreas Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: interim analysis found the study drug to be ineffective
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dana Cardin, MD, Assistant Professor of Medicine; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 1016; NCI-2010-02123
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-06

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — STA 9090; Phantoms, Imaging; Magnetic Resonance Spectroscopy; X-Rays; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- STA-9090 (Experimental): Patients receive Hsp90 inhibitor STA-9090 IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: STA-9090; Radiation: Radiologic imaging; Procedure: blood draw

INTERVENTIONS:
Drug: STA-9090 — Given IV
Radiation: Radiologic imaging — radiologic modalities used to evaluate response to treatment
  Other Names: computerized tomographic (CT) scan; magnetic resonance imaging (MRI); chest x-ray
Procedure: blood draw — Venous blood will be drawn from those patients who give consent. Serum will be used to look for biomarkers predictive of response

SUMMARY:
RATIONALE: Heat shock protein (HSP)90 inhibitor STA-9090 may stop the growth of tumor cells by blocking some of the proteins needed for cell growth. PURPOSE: This phase II trial is studying how well hsp90 inhibitor STA-9090 works as second- or third-line therapy for the treatment of patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To measure the 8-week disease control (CR + PR + SD) rate of therapy with STA-9090 in patients with metastatic pancreas cancer who have failed (either progressed or did not tolerate) one or two lines of prior therapy. SECONDARY OBJECTIVES: I. To determine response rate (by RECIST criteria v1.1). II. To determine overall survival. III. To evaluate the safety and toxicity profile in this patient population. TERTIARY OBJECTIVES: I. We will obtain from all patients blood samples pre and post therapy (after 1 week of therapy) and isolate serum for interrogation for a variety of biomarkers (eg AKT, Stat3, Caspase 3). OUTLINE: Patients receive Hsp90 inhibitor STA-9090 intravenous (IV) over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Microscopic confirmation of a diagnosis of metastatic adenocarcinoma (pathology may be from either the primary tumor or metastatic lesion) or poorly differentiated carcinoma of the pancreas s/p 1 or 2 prior chemotherapy regimens for metastatic disease (excluding neuroendocrine tumors, periampullary tumors and cystadenocarcinoma)
* Patients who received adjuvant or neoadjuvant therapy will be eligible if they have progressed within 6 months of completing therapy and have not received a metastatic regimen or if they progressed > 6 months after completing therapy and have received 1-2 lines of therapy for metastatic disease
* Measurable disease by RECIST criteria
* ECOG PS 0 or 1
* Life expectancy of at least 12 weeks
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine =< 2.0 mg/dl
* Total bilirubin =< 2.0 mg/dl
* AST and ALT =< 2.5 x ULN in absence of liver metastasis; =< 5 x ULN in presence of liver metastasis
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of therapy
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent; a signed informed consent must be obtained prior to any study-specific procedures

Exclusion Criteria:

* Primary brain tumors or active brain metastases; however, patients with a history of CNS metastases will be eligible if they have been treated and are stable for 4 weeks after completion of treatment, with image documentation required, and must be either off steroids or on a stable dose of steroids for a minimum of 2 weeks prior to enrollment
* History of stroke within 6 months of treatment or other significant neurological limitations
* History of or current coronary artery disease, myocardial infarction, angina pectoris, angioplasty of coronary bypass surgery
* History of or current uncontrolled dysrhythmias, or requirement for antiarrhythmic medications, or Grade 2 or greater left bundle branch block
* New York Heart Association class II/III/IV congestive heart failure with a history of dyspnea, orthopnea or edema that required current treatment with angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, beta-blockers or diuretics
* Current or prior radiation therapy to the left hemithorax
* Major surgery within 4 weeks prior to entering the study
* Poor venous access for study drug administration or would require a peripheral or central indwelling catheter for study drug administration; study drug administration via indwelling catheters is prohibited at this time
* Use of any investigational agents within 4 weeks prior to entering the study
* History of severe allergic reactions to excipients (e.g., Polyethylene glycol 300 and Polysorbate 80), including severe hypersensitivity reactions defined as >= Grade 3 based on NCI CTCAE version 4.0
* Treatment with chronic immunosuppressants (e.g., cyclosporine following transplantation or systemic steroids for treatment of autoimmune disease), however, patients may receive steroids for stable CNS metastases as described in exclusion criterion 1
* Uncontrolled intercurrent illness including, but not limited to, human immunodeficiency virus (HIV)-positive patients receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study
* Ventricular ejection fraction (Ef) =< 55%
* Baseline QTc > 470 msec or previous history of QT prolongation while taking other medications
* Patients who received more than two lines of prior therapy for metastatic disease, neoadjuvant or post-op adjuvant therapy is not considered one line of therapy as long as there was > 6 months of disease-free interval
* Pregnant or breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Cardin, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - The Jones Clinic, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened in December 2010 and ran to April 2013
Pre-assignment Details: Seventeen patients consented to this study, 2 were determined ineligible to participate
Groups:
- STA-9090: 175 mg/m2 STA-9090 intravenously (IV) over 1 hour once a week for 3 weeks (Day 1, Day 8 and Day 15), followed by a 1 week dose-free interval. The 4-week treatment cycle continues to disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | STA-9090
Started | 15
Completed | 0
Not Completed | 15
Not completed — Disease progression | 9
Not completed — Toxicity | 2
Not completed — Withdrew after beginning treatment | 4

BASELINE CHARACTERISTICS:
Arm/Group | STA-9090
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 65 (11) [33 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate
Description: Per RECIST criteria v. 1.0: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions, and progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions. Disease control is defined as CR + PR + SD after 8 weeks of therapy.
Time Frame: at 8 weeks from the start of therapy
Population: Patients who received treatment and who were available for determination of response.
Measure: Number; unit: percentage of participants
Arm/Group | STA-9090
Number analyzed (Participants) | 11
percentage of participants | 21

2. Secondary Outcome: Best Response
Description: Number of patients in each response category, per RECIST v1.1, summarized as follows for target lesion criteria (see RECIST v1.1 for additional details): complete response (CR),disappearance of target lesions; partial response (PR), >=30% decrease in sum of longest diameter of target lesions; progressive disease (PD), >=20% increase in sum of LD of target lesions or appearance of new lesions; stable disease (SD), insufficient change in target lesions or new lesions to qualify as either PD or SD. Patients are categorized according to the best response achieved prior to occurrence of progressive disease, where best response hierarchy is CR>PR>SD>PD.
Time Frame: On-treatment date, to date of disease progression (assessed up to 1 year)
Population: All patients with best overall response data; patients are excluded if best overall response data is missing or if the patient is non-evaluable for best overall response.
Measure: Number; unit: participants
Arm/Group | STA-9090
Number analyzed (Participants) | 15
participants
  Complete response | 0
  Partial response | 0
  Stable disease | 3
  Progressive disease | 8
  Not Assessed | 3
  Not Evaluable | 1

3. Secondary Outcome: Overall Survival
Description: Estimated probable duration of life from on-study date to date of death from any cause, using the Kaplan-Meier method with censoring (see analysis population description for additional details)
Time Frame: study entry to date of death or last date known alive (assessed over 2.5 yrs)
Population: All patients are included in the analysis on intention-totreat basis. Analysis is by Kaplan-Meier method, where death is an event, with censoring for non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | STA-9090
Number analyzed (Participants) | 15
days | 125 [45 to 148]

4. Secondary Outcome: Number of Patients With Each Worst Grade Toxicity
Description: Count of patients according to the worst-grade toxicity experienced by each, where worst-grade toxicity is per NCI common toxicity criteria: grade 1, mild; grade 2, moderate; grade 3, severe; grade 4, life-threatening; grade 5, death
Time Frame: On study date to 30 days following final dose of study drug
Population: Total number of patients reported with any toxicity related to study treatment. One patient withdrew before treatment. One patient did not have a toxicity related to study drug or therapy.
Measure: Number; unit: participants
Arm/Group | STA-9090
Number analyzed (Participants) | 13
participants
  Patients with worst grade toxicity 1 | 0
  Patients with worst grade toxicity 2 | 5
  Patients with worst grade toxicity 3 | 8
  Patients with worst grade toxicity 4 | 0
  Patients with worst grade toxicity 5 | 0

5. Other Pre Specified Outcome: Biomarker Evaluation
Description: Serum will be tested for biomarkers that may be predictive of response, optional per patient consent.
Time Frame: Pre-treatment and 1 week post-treatment
Population: The study's interim analysis found the study drug to be ineffective. The study was terminated. No biomarkers were performed or analyzed.
Arm/Group | STA-9090
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- STA-9090: 175 mg/m2 STA-9090 IV over 1 hour once a week for 3 weeks, followed by a 1 week dose-free interval. The 4-week treatment cycle continues to disease progression.
Arm/Group | STA-9090
Serious Adverse Events (participants affected / at risk) | 9/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STA-9090 (N=14)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
acute kidney injury (Renal and urinary disorders) | 1 (1)
alanine aminotransferase increased (Investigations) | 1 (1)
alkaline phosphatase increased (Investigations) | 1 (1)
ascites (Gastrointestinal disorders) | 1 (1)
aspartate aminotransferase increased (Investigations) | 1 (1)
biliary tract infection-cholangitis (Hepatobiliary disorders) | 1 (1)
chills (General disorders) | 1 (1)
confusion (Psychiatric disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 2 (2)
dyspnea (Reproductive system and breast disorders) | 1 (1)
failure to thrive (General disorders) | 1 (1)
gastric perforation (Gastrointestinal disorders) | 1 (1)
hepatic failure (Hepatobiliary disorders) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
malaise (General disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 3 (3)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
renal calculi (Renal and urinary disorders) | 1 (1)
thromboembolic event (Vascular disorders) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 2 (2)
blood bilirubin increased (Hepatobiliary disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STA-9090 (N=14)
abdominal pain (Gastrointestinal disorders) | 9 (16)
diarrhea (Gastrointestinal disorders) | 8 (25)
constipation (Gastrointestinal disorders) | 7 (10)
nausea (Gastrointestinal disorders) | 6 (16)
vomiting (Gastrointestinal disorders) | 3 (10)
flatulence (Gastrointestinal disorders) | 2 (2)
gastrointestinal disorders-other (Gastrointestinal disorders) | 2 (2)
ascites (Gastrointestinal disorders) | 1 (1)
bloating (Gastrointestinal disorders) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 1 (2)
esophageal pain (Gastrointestinal disorders) | 1 (1)
hemorrhoids (Gastrointestinal disorders) | 1 (1)
rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 8 (16)
hypokalemia (Metabolism and nutrition disorders) | 6 (8)
anorexia (Metabolism and nutrition disorders) | 4 (4)
dehydration (Metabolism and nutrition disorders) | 4 (4)
hyperglycemia (Metabolism and nutrition disorders) | 4 (9)
hypoalbuminemia (Metabolism and nutrition disorders) | 4 (10)
hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
metabolism and nutrition disorders-other (Metabolism and nutrition disorders) | 1 (2)
alkaline phosphatase increased (Investigations) | 8 (13)
alanine aminotransferase increased (Investigations) | 6 (9)
aspartate aminotransferase increased (Investigations) | 5 (8)
lymphocyte count decreased (Blood and lymphatic system disorders) | 5 (8)
blood bilirubin increased (Hepatobiliary disorders) | 4 (7)
platelet count decreased (Blood and lymphatic system disorders) | 4 (4)
weight loss (Metabolism and nutrition disorders) | 3 (4)
creatinine increased (Investigations) | 1 (1)
fatigue (General disorders) | 9 (18)
edema limbs (General disorders) | 3 (4)
pain (General disorders) | 2 (2)
chills (General disorders) | 1 (1)
edema face (General disorders) | 1 (1)
general disorders-other (General disorders) | 1 (2)
anemia (Blood and lymphatic system disorders) | 7 (11)
blood and lymphatic system disorders-other (Blood and lymphatic system disorders) | 1 (1)
dysgeusia (Nervous system disorders) | 2 (2)
headache (Nervous system disorders) | 2 (2)
dizziness (Nervous system disorders) | 1 (1)
nervous system disorders-other (Nervous system disorders) | 1 (1)
paresthesia (Nervous system disorders) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
tremor (Nervous system disorders) | 1 (1)
depression (Psychiatric disorders) | 3 (4)
insomnia (Psychiatric disorders) | 2 (3)
confusion (Psychiatric disorders) | 1 (2)
psychosis (Psychiatric disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
musculoskeletal and connective tissue disorder-other (Musculoskeletal and connective tissue disorders) | 1 (1)
pain-extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
cardiac disorder-other (Cardiac disorders) | 1 (1)
sinus bradycardia (Cardiac disorders) | 1 (2)
sinus tachycardia (Cardiac disorders) | 1 (1)
bruising (Injury, poisoning and procedural complications) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1)
renal and urinary disorder-other (Renal and urinary disorders) | 2 (3)
urinary frequency (Renal and urinary disorders) | 1 (1)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
hypotension (Vascular disorders) | 2 (2)
lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
irritability (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes